CLINICAL TRIAL: NCT06713265
Title: Study of the Link Between Freezing of Gait and Oropharyngeal Freezing in Parkinson's Patients
Acronym: Freez in park
Status: Recruiting | Type: Observational
Sponsor: Hopital La Musse (Other)
Responsible Party: Sponsor
Other Study IDs: 2024-A01781-46
Record Dates: First submitted 2024-11-27; First posted 2024-12-03 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-09

CONDITIONS: Parkinson's Disease; Dysphagia; Swallowing Disorder; Freezing of Gait; Oropharyngeal Disease; Gait Disorders
Keywords: Parkinson's Disease; Dysphagia; Swallowing disorder; Freezing of gait; oropharyngeal freezing; Gait
MeSH Terms: conditions — Parkinson Disease; Deglutition Disorders; Mobility Limitation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- With freezing of gait: During patient enrollment, the following assessments will be conducted:
  * The Unified Parkinson's Disease Rating Scale (UPDRS);
  * Timed Up & Go (TUG) Test;
  * New Freezing of Gait Questionnaire (NFOG-Q);
  * BAASTA Battery;
  * Clinical swallowing assessment. All assessments will be conducted during the patient's OFF phase.
  At the end of the motor assessment (NFOG-Q and TUG), the patients will be divided into two groups: the first group will consist of patients exhibiting freezing of gait, while the second group will consist of those not presenting freezing. The procedure for the assessments will remain the same for both groups.
  If, during the clinical speech therapy swallowing assessment, signs indicative of swallowing disorders are detected, the patient will be referred for a pharyngography to specify the nature of these disorders.
- Without freezing of gait: During patient enrollment, the following assessments will be conducted:
  * The Unified Parkinson's Disease Rating Scale (UPDRS);
  * Timed Up & Go (TUG) Test;
  * New Freezing of Gait Questionnaire (NFOG-Q);
  * BAASTA Battery;
  * Clinical swallowing assessment. All assessments will be conducted during the patient's OFF phase.
  At the end of the motor assessment (NFOG-Q and TUG), the patients will be divided into two groups: the first group will consist of patients exhibiting freezing of gait, while the second group will consist of those not presenting freezing. The procedure for the assessments will remain the same for both groups.
  If, during the clinical speech therapy swallowing assessment, signs indicative of swallowing disorders are detected, the patient will be referred for a pharyngography to specify the nature of these disorders.

SUMMARY:
Parkinson's Disease: Study of the Link Between Gait Freezing and Oropharyngeal Freezing Parkinson's disease is the second most common neurodegenerative disorder worldwide. Parkinsonian dysphagia is a frequently encountered disorder in this condition, affecting all phases of swallowing: oral, pharyngeal, and esophageal. This dysphagia can occur at any stage of the disease. While most swallowing difficulties develop in the advanced stages of Parkinson's disease, they can also appear early on and are often underdiagnosed. The prevalence of swallowing disorders in Parkinson's disease is estimated to range from 40% to 80%, with this variability explained by the significant differences in the precision of swallowing evaluations conducted and the fact that dysphagia is still too frequently underdiagnosed. Yet, dysphagia is the leading cause of mortality in Parkinson's patients.

Dysphagia can negatively affect patients' quality of life. It leads to difficulties during oral intake (food, liquids, and medications), weight loss, dehydration, malnutrition, and limitations in social activities. Depression is frequently associated with reduced quality of life in Parkinson's patients with swallowing disorders. Moreover, aspiration pneumonia due to mis-swallowing is one of the primary reasons for hospitalization in Parkinson's patients, potentially leading to severe complications and, at times, death.

Oropharyngeal freezing, also called oral festination, is an involuntary, repetitive anteroposterior movement of the tongue against the soft palate performed before transferring the food bolus to the pharynx. This movement is also observed during multiple swallows. This phenomenon is more frequent in dysphagic Parkinson's patients, yet its impact on swallowing dynamics remains poorly understood. Oropharyngeal freezing has been observed in approximately 40% to 75% of Parkinson's patients during videofluoroscopic swallow studies, also known as swallowing pharyngography. Oropharyngeal freezing inhibits the initiation of swallowing, keeping the airway open and leading to tracheal aspiration of residues. Some fragments then slide into the valleculae and pyriform sinuses. Thus, oropharyngeal freezing exacerbates pharyngeal phase incoordination, increasing the risk of aspiration pneumonia. Therefore, addressing this swallowing disorder is essential.

Oropharyngeal freezing is intrinsically rhythmic. While limited studies have been conducted on the topic, they agree that gait freezing (difficulty initiating walking, stopping in response to obstacles, or circumventing them) and oropharyngeal freezing share common pathophysiological mechanisms. Gait freezing is not limited to deficits in the locomotor network but is part of a broader deficit affecting spatiotemporal coordination in various tasks, similar to oropharyngeal freezing.

It is, therefore, crucial to detect this oral phase swallowing disorder as early as possible, enabling tailored early intervention that helps patients maintain their swallowing abilities for as long as possible and prevents complications mentioned earlier. Since gait freezing is diagnosed much earlier and more systematically, it would be interesting to investigate whether there is a correlation between the presence of gait freezing and oropharyngeal freezing in these patients. This could guide patients with gait freezing toward early speech-language assessments to evaluate the presence of oropharyngeal freezing.

The objectives of the study are examine the prevalence of oropharyngeal freezing in Parkinson's patients. Based on the results obtained from the NFOG-Q (New Freezing of Gait Questionnaire), two groups will be formed: The first group will consist of patients exhibiting gait freezing. The second group will consist of patients without gait freezing. The secondary objectives of the study are examine the common characteristics between these two types of freezing (gait and oropharyngeal). To assess the sensitivity and reliability of the NFOG-Q in detecting oropharyngeal freezing.To determine the prevalence of oropharyngeal freezing based on the score obtained on the UPDRS (Unified Parkinson's Disease Rating Scale). To analyze the link between patients' rhythmic abilities and the presence or absence of one or both types of freezing.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of idiopathic Parkinson's disease established by a neurologist;
* Patient affiliated with the social security system;
* Patient aged over 18 years.

Exclusion Criteria:

* Patients under legal protection measures;
* Neurological history that could be the cause of a swallowing disorder (e.g., stroke) or a history of ENT cancer;
* Patient with a gastrostomy without oral intake;
* Pregnant women or those suspected of being pregnant;
* Minor patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The chosen study population consists of patients with idiopathic Parkinson's disease.
Sampling Method: Probability Sample
Enrollment: 66 (Estimated)
Dates: Start 2024-10-04 (Actual); Primary Completion 2025-10-31 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
The judgment of the presence or absence of oropharyngeal freezing during a pharyngography in the OFF phase of an idiopathic Parkinson's disease patient. | At the enrollement
  Pharyngography is a swallowing examination that allows for recording films of the patient's swallowing using a radiological device. The radiology device will be positioned at the patient's neck and will record these sequences. Once the device is in place, the patient will swallow bites of varying thickness. For all swallowing actions, barium will be used, which is a radiopaque, white substance with a slightly mentholated taste.

SECONDARY OUTCOMES:
The objective assessment of the severity, fluctuation, and progression of clinical symptoms, as well as their impact on the patient's daily life. | At the enrollement
  The Unified Parkinson's Disease Rating Scale (UPDRS) is a composite measurement tool that combines several evaluation scales and is organized into six sections. It is a multidimensional scale that allows for an objective assessment of the severity, fluctuations, and progression of clinical symptoms, as well as their impact on the patient's daily life.
  The first section evaluates the patient's mental, behavioral, and mood state. The second section allows for a self-assessment of activities of daily living. The third section assesses motor functions, while the fourth section evaluates treatment complications over the week prior to the examination. The fifth section involves the administration of the Hoehn and Yahr scale, which classifies patients into five main stages based on the severity of their condition. The final section is the Schwab and England quality of life scale, which evaluates the patient's ability to perform activities of daily living in terms of speed and autonomy.
Assessment of gait freezing | At the enrollement
  The New Freezing of Gait Questionnaire (NFOG-Q) is a 9-item questionnaire excluding patients with no freezing in item 1, duration and frequency of freezing in items 2 to 6, and the impact of freezing on daily activities in items 7 to 9). The concurrent validity is poor when compared to the freezing time in a TUG test and the number of freezing events that occurred. The reliability and internal consistency are good. Video assistance may improve scoring.
Assessment of gait freezing 2 | At the enrollement
  The Timed Up and Go (TUG) test is a simple test conducted during a consultation: the subject, seated on a chair, must stand, walk 3 meters, turn around, and return to sit. The score is given by the time in seconds. The test is normal if the time is less than 14 seconds (or 20 seconds according to some publications). The TUG test has good reproducibility over time and between observers. Its sensitivity is 87%, and its specificity is 87%.
Rhythm assessment | At the enrollement
  The BAASTA Battery is a series of tests on a touchscreen tablet that assess rhythmic perceptual and sensorimotor abilities. It is used to detect deficits in rhythmic abilities through patented measurement methods and is designed for researchers and healthcare providers to assess the motor synchronization of their subjects/patients. They perform a series of exercises to evaluate their rhythmic abilities, such as tapping in time with sounds, music, and detecting isochrony errors.
Assessment of swallowing disorders | At the enrollement
  The Modified Barium Swallow Impairment Profile (MBSImP) is a standardized protocol for pharyngography to interpret and communicate swallowing disorders in a specific, consistent, precise, and objective manner.
Assessing functional swallowing ability over time | At the enrollement
  The Functional Oral Intake Scale (FOIS) is a scale used to document any changes in a patient's diet, reflecting the evolution of their functional swallowing abilities over time. Level 1 corresponds to "nothing by mouth," and level 7 corresponds to a "complete oral diet without restriction." This scale will be used during the clinical speech therapy assessment.
Assessming of the severity of aspiration events | At the enrollement
  The Penetration Aspiration Scale (PAS) evaluates the severity of aspiration events. It is an 8-point scale, where score 1 indicates normal swallowing, and score 8 represents the most severe level, corresponding to silent aspiration. This scale will be used during nasofibroscopy and pharyngography exams.
Quantitative assessment of the effectiveness of solid food ingestion | At the enrollement
  The Test of Masticating and Swallowing Solids (TOMASS) allows for a quantitative assessment of the effectiveness of solid food ingestion. The patient is asked to eat a Tuc cracker as quickly and comfortably as possible and to state their name after the last swallow. The goal is to quantitatively evaluate the chewing and swallowing of a solid bolus. The examiner records the number of bites, chewing cycles, swallows, and total time. Norms are established based on age and gender, as these are considered influential factors on chewing. This test will be conducted during the clinical speech therapy assessment.
Quantitative evaluation of the effectiveness of liquid bolus ingestion | At the enrollement
  The Waster Swallowing Test (TWST) provides a quantitative evaluation of the effectiveness of liquid bolus ingestion. The patient is asked to drink a glass of water (150 mL for patients under 75 years old, and 100 mL for those over 75 years old) as quickly and comfortably as possible. The goal is to quantitatively evaluate liquid swallowing. The number of swallows and the total ingestion time are recorded. This test will be conducted during the clinical speech therapy assessment.
Detection of clinical signs of dysphagia, including silent aspirations | At the enrollement
  The Volume-Viscosity Swallow Test (V-VST) offers a quick, safe, and accurate diagnostic test to detect clinical signs of dysphagia, including silent aspirations. The test is detailed and easy to use, with good sensitivity (88.2%) and specificity (64.7%). The V-VST protocol includes three texture tests in this order: nectar, paste, and liquid. The liquid is colored with either mint or grenadine syrup, based on patient preference, to improve visual and taste appeal. Each texture is tested in three different volumes (5, 10, 20 mL) using both a spoon and a glass, while monitoring oxygen saturation with a fingertip pulse oximeter. Swallowing disorders are divided into two main categories: propulsion disorders and airway protection disorders.
Assessment of the quality of life of patients with oropharyngeal dysphagia | At the enrollement
  The Swallowing Quality of Life (SWAL-QOL) is a 44-item questionnaire that addresses 10 concepts related to the quality of life of patients with oropharyngeal dysphagia. Each concept corresponds to a subscale: the burden of swallowing difficulties, meal duration, desire to eat, food choices, communication, fear, mental health, social impact, fatigue, and sleep. Each item is rated on a 5-point scale, and the total score is calculated, with a maximum score of 100. The lower the score, the worse the quality of life. This test will be conducted during the clinical speech therapy assessment.

CONTACTS AND LOCATIONS:
Overall Officials: Héloïse BAILLET, PhD, Principal Investigator — Hôpital La Musse; Eric VERIN, PU-PH, Study Director — CHU Rouen, GRHVN Laboratory
Locations (1):
- Hôpital La Musse, Saint-Sébastien-de-Morsent, France

IPD SHARING:
Plan to Share IPD: Undecided